CLINICAL TRIAL: NCT01611285
Title: Uphold Versus Robotic Surgery for Pelvic Prolapse Repair: A Decision Analytic Approach
Status: Completed | Type: Observational
Sponsor: Atlantic Health System (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: R10-04-002
Record Dates: First submitted 2012-05-30; First posted 2012-06-04 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Pelvic Organ Prolapse
Keywords: UPHOLD; robotic surgery; decision analysis; FDA; decision node; outcome node
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Robotic Sacrocolpopexy patients: Patients who underwent Robotic Sacrocolpopexy to treat pelvic organ prolapse between 2009 and 2010
- UPHOLD patients: Patients who underwent the UPHOLD procedure to treat pelvic organ prolapse from 2009-2010.

SUMMARY:
Within the general objective of investigating optimal medical techniques for pelvic prolapse repair, this study proposes to: (1) test the hypothesis that the UPHOLD procedure is more cost effective than robotic surgery for pelvic prolapse repair (2)using formal decision analysis as the comparative strategy

DETAILED DESCRIPTION:
The cumulative incidence of pelvic organ prolapse was approximately 2% in 2001. Given the aging demographics in the U.S., the incidence of prolapse is projected to increase to 30% or more for women aged 60 years and older and become of greater concern to both patients and physicians. The demand for gynecologic services is predicted to increase by more than 45% in the next ten years. Prolapse is related to childbirth, aging, defects in collagen, and smooth muscle structure and strength. Etiology includes intra-abdominal pressure from obesity, with obesity becoming an ever increasing factor in the US.

Treatment Choice of Patients:

Patients choose between pessary, surgery, and expectant management based on: age, prior prolapse surgery, preoperative pelvic pain scores, and pelvic organ prolapse severity. These are difficult decisions for patients.

When it comes to choosing between destinctive interventions with subtle advantages and disadvantages, patients typically want to hear their physician's views of the scientific merits of each procedure. Informed consent becomes extremely difficult when issues of cost-effectiveness are at hand. Thus, the proposed project.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Underwent either UPHOLD procedure or Robotic Surgery for Pelvic Organ prolapse

Exclusion Criteria:

* Other vaginal procedure to correct prolapse

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients who underwent either robotic surgery or the UPHOLD procedure to treat pelvic organ prolapse from 2009-2010
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Surgical cure versus failure of prolapse repair | within 12 months of patients surgery
  Incidence of recurrance of pelvic organ prolapse within 12 months of either robotic sacrocolpopexy or the UPHOLD procedure

SECONDARY OUTCOMES:
Financial costs of outcomes | within 12 months of patients surgery
  Financial costs that will incur to produce the primary outcomes- success or failure. When the two outcomes are considered together, we have "cost effectiveness"

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Culligan, MD FACOG FACS, Principal Investigator — Atlantic Health System
Locations (1):
- Atlantic Health System Department of Urogynecology, Morristown, New Jersey, United States